CLINICAL TRIAL: NCT01228240
Title: The Efficacy of Metformin Produced by Pars Mino Co in Comparison With Canadian Apotex Co.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zanjan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Majid Valizadeh, Professor, Zanjan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 19/3-3/2073
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2 AND Metformin
Keywords: Diabetes mellitus, type 2, Metformin, Generic, Efficacy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Metformin, Apo-metformin (Experimental): Participants under treatment with non-generic Metformin (manufactured by Apotex Canada).
  Interventions: Drug: Metformin
- Metformin, Pars Minoo (Active Comparator): Participants under treatment with generic Metformin (manufactured by Pars Minoo).
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Background: Metformin is usually using for glycemic control in type 2 diabetes mellitus. Different pharmaceutical types of metformin are available. As a clinical trial, we compared the efficacy and complications of metformin produced by "Pars Mino pharmaceutical company, Iran" with "Apotex pharmaceutical company, Canada", in type 2 diabetic patients.

Method: 18 eligible women with type 2 diabetes were given metformin "Pars Mino" or "Apotex" (500 mg twice a day) each for 6 weeks period in a randomized, double blind, crossover study. These two groups randomly under treatment with generic metformin (manufactured by Pars Mino company) or non-generic (manufactured by Apotex Canada). After 2 weeks washout period another 6 weeks period with another Brand of metformin was prescribed. FBS, HbA1C, lipid profile (Cholesterol, TG, HDL, and LDL), weight, and BMI were assessed before and after each treatment phase. The results were compared with each other by paired sample T-test, Independent sample T-test.

ELIGIBILITY:
Inclusion Criteria:

* Mild hyperglycemia, no contraindication for metformin, poor controlled diabetes

Exclusion Criteria:

* Creatinine more than 1.5, severe organ damage

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)